CLINICAL TRIAL: NCT01977495
Title: Testing Enrollment Methods on Participation in Behavioral Economic Interventions for Diabetes Care: A Randomized Controlled Pilot Study
Brief Title: Take Charge of Your Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Jaya Aysola, Principal Investigator, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 818810
Record Dates: First submitted 2013-10-24; First posted 2013-11-06 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes; Hypertension
Keywords: Diabetes; Enrollment methods; Behavioral Economic Intervention; Opt-in Enrollment; Opt-out Enrollment; lottery; financial incentives
MeSH Terms: conditions — Diabetes Mellitus; Hypertension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Opt-in Enrollment (Active Comparator): Opt-in enrollment: patient will be sent a recruitment letter, in which they must call the study team to take part in the study. During that call, the study team will schedule the participant for an intake visit.
  Interventions: Behavioral: Financial Incentive: Fixed Lottery
- Opt-out enrollment (Active Comparator): Opt-out enrollment: patient will be sent a letter communicating to them that they have been enrolled into a research program at their doctor's office. After 10 days, the study team will contact the opt-out participants to schedule an intake visit.
  Interventions: Behavioral: Financial Incentive: Fixed Lottery

INTERVENTIONS:
Behavioral: Financial Incentive: Fixed Lottery — Every day of the 91 day intervention period participants will be asked to use each of their biometric devices. A daily lottery will be conducted automatically by the study website. Participants must use each of their two devices daily to be eligible for the lottery the following day. Winning lottery numbers will be identified by a fixed-position match between the automatically generated winning number and a participant ID number, which each participant will pick at enrollment.

SUMMARY:
The investigator plans to assess enrollment rates among two different enrollment methods, while providing a behavioral economic intervention to enhance the uptake of home-health monitoring devices to lower hemoglobin A1C among patients with uncontrolled diabetes. The study is focusing on enrollment methods since the standard randomized control trial only reaches 15% of the population. The study is seeking to understand the effectiveness of a behavioral intervention, when rolled out in a larger population.

ELIGIBILITY:
Inclusion Criteria:

1. Adults between 18 and 80 years of age
2. Primary care patients at the Division of General Internal Medicine clinics at the University of Pennsylvania
3. Hemoglobin A1c measured within the last 8 weeks greater than 8.0% OR no measured Hemoglobin A1C measured in the last two years
4. A confirmed diabetes diagnosis
5. Planning to stay in area for study duration (6 months)
6. Can understand and communicate fluently in English

Exclusion Criteria:

1. Unable to read and give consent
2. Suffer from an uncontrolled psychiatric disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-12; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Enrollment and participation rates | End of study- 6 months after enrollment
  The primary objective is to obtain preliminary evidence regarding whether or not patients opt-into a research study, as opposed to enrolling by default, will affect participation in the program and the effectiveness of the intervention, among high-risk patients. The primary outcome is to measure enrollment rates. The investigators will also measure participation in the program through device usage.

SECONDARY OUTCOMES:
Uptake of Device Usage | End of study- 6 months after enrollment
  Assess the effect of financial incentives on the use of home health monitoring devices among high-risk patients

OTHER OUTCOMES:
Change in Hemoglobin A1c | End of study- 6 months after enrollment
  Assess how regular use of home-based health monitoring devices affects clinical outcomes, such as Hemoglobin A1C

CONTACTS AND LOCATIONS:
Overall Officials: Jaya Aysola, MD, MPH, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States